CLINICAL TRIAL: NCT01245985
Title: Induction Chemotherapy With TPF Followed by Radioimmunotherapy With Cetuximab and Intensity Modulated Radiotherapy (IMRT) Plus Carbon Ion Boost for Locally Advanced Tumors of the Oro-, Hypopharynx and Larynx: TPF-C-HIT
Brief Title: TPF Followed by Cetuximab and IMRT Plus Carbon Ion Boost for Locally Advanced Head and Neck Tumors
Acronym: TPF-C-HIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment (only 8 patients recruited and treated until 12/2012)
Sponsor: Heidelberg University (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: PD Dr. Marc Muenter, Dept of Radiation Oncology, University of Heidelberg, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPF-C-HIT
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN): Oro-, Hypopharyngeal and Laryngeal Cancer
Keywords: SCCHN; squamous cell carcinoma of the head and neck; oropharyngeal carcinoma; hypopharyngeal carcinoma; laryngeal carcinoma
MeSH Terms: conditions — Laryngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment arm (Experimental): patients receive induction chemotherapy with TPF for a maximum of 3 cycles followed by radioimmunotherapy with cetuximab as intensity-modulated radiotherapy (IMRT) plus carbon ion boost
  Interventions: Radiation: carbon ion boost

INTERVENTIONS:
Radiation: carbon ion boost — patients receive induction chemotherapy with TPF for a maximum of 3 cycles followed by radioimmunotherapy with cetuximab as intensity-modulated radiotherapy (IMRT) plus carbon ion boost

SUMMARY:
TPF-C-HIT investigates the combination of induction chemotherapy with TPF followed by radioimmunotherapy with cetuximab and IMRT plus carbon ion boost with regard to efficacy and toxicity of the combination regimen.

DETAILED DESCRIPTION:
TPF-C-HIT is a prospective, monocentric phase II trial efficacy, as measured by control and survival rates, as well as toxicity (acute and late effects) of the combined treatment with TPF-induction followed by radioimmunotherapy with the EGFR-antibody cetuximab and carbon ion boost in locally advanced squamous cell carcinoma of the head and neck (SCCHN). As long-term local control remains a therapeutic challenge in advanced head and neck cancer, locoregional control was chosen as the primary endpoint. Secondary endpoints are survival rates (disease-free survival, PFS, OS), acute and late radiation effects as well as adverse events. For development of prognostic markers, proteomic and genomic analyses are also included in the secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent,
* Age of 18 to 70 years,
* Life expectancy of at least 6 month,
* Ability of subject to understand character and individual consequences of clinical trial,
* Histologically confirmed locally advanced (stage III or IV), non-metastatic squamous cell carcinoma of oro-, hypopharynx and larynx (T2-4, any N, M0),
* Oral cavity or oro- , hypopharynx or laynx as the primary tumor site,
* At least one uni-measurable lesion according to the RECIST criteria, Karnofsky Performances Status > 70%,
* Adequate bone marrow function: neutrophils > 1.5 x 109/L, platelets > 100 x 109/L, hemoglobin > 10.0 g/dL,
* Adequate liver function: Bilirubin < 1.5 mg/dL, SGOT, SGPT < 3 x ULN, GGT < 5 x ULN,
* Adequate renal function: GFR> 70 ml/min,
* Negative serum/urine Beta-HCG test in women of childbearing potential,
* Women of childbearing potential: willingness to use effective contraceptive method, defined as the concomitant use of either an intrauterine pessary (IUP) or contraceptive pill and in both cases, condoms for the treatment duration and 2 months thereafter. Women of non-childbearing potiential are those who are post-menopausal for at least 1 year or sterilized,
* Men of procreative potential: willingness for effective prevention of procreation, defined as a use of condoms and a use of either an intrauterine pessary (IUP) or a contraceptive pill by his partner for the treatment duration and 2 months thereafter,
* Subject's consent to collect blood and/or tumor tissue samples for proteomics and genomics. If a patient does not consent, no samples for proteomics and genomics will be taken. Nonetheles, he/she may be enroled in the study

Exclusion Criteria:

* Previous systemic chemotherapy, radiotherapy or surgery for carcinoma of the head, neck and larynx,
* Nasopharyngeal Carcinoma,
* Prior exposure to EGFR pathway targeting therapy,
* Evidence of distant metastases.
* Other serious illness or medical conditions:
* Unstable cardiac disease despite treatment, congestive heart failure NYHA grade 3 and 4,
* Significant neurologic or psychiatric disorders including dementia or seizures,
* Active disseminated intravascular coagulation,
* Other serious underlying medical conditions which in the opinion of investigator could impair the ability of the patient to participate in the study,
* Symptomatic peripheral neuropathy Common Toxicity Criteria (CTC) grade 2 or higher,
* ototoxicity CTC grade 2 or higher, except if due to trauma or mechanical impairment due to tumor mass,
* Participation in other interventional trial within the last 30 days§§,
* Surgery within the last 30 days,
* Known allergic/hypersensitivity reaction to any drugs scheduled for the study treatment,
* Women: pregnant or breast-feeding,
* Known drug abuse,
* Other previous malignancy within 5 years, with exception of a history of a previous, adequately treated, basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix,
* Legal incapacity or limited legal capacity,
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Local-Regional Control (LRC) | 12 months
  The primary endpoint of the study is the Local-Regional Control (LRC) at 1 year

SECONDARY OUTCOMES:
disease-free survival (DFS) | 12 months
progression-free survival (PFS) | 12 months
overall survival (OS) | 12 months
acute radiation effects | 6 weeks post completion of radiotherapy
late radiation effects | 12 months
adverse events | 12 months
  includes any adverse events attributable to the combined treatment not otherwise specified
proteomic and genomic analyses | 6 measuring points: days 50, 64, 73, 106 of treatment; 6 weeks post completion of radioimmunotherapy; 3 months post completion of radioimmunotherapy
  proteomic and genomic analyses designed to investigate changes during therapy, therefore analyses are carried out at 6 measuring points: days 50, 64, 73, 106 of treatment; 6 weeks post completion of radioimmunotherapy; 3 months post completion of radioimmunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc W Muenter, MD, Principal Investigator — Heidelberg University
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, Heidelberg, Germany